CLINICAL TRIAL: NCT04640402
Title: A Single-center, Randomized, Double-Blinded, Placebo-Controlled, Phase Ⅱ Clinical Trial of Recombinant COVID-19 Vaccine (Sf9 Cells), in the Subjects From Healthy Aged 18 Years and Above
Brief Title: A Phase Ⅱ Clinical Trial of Recombinant Corona Virus Disease-19 (COVID-19) Vaccine (Sf9 Cells)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT099
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Safety; Immunogenicity; COVID-19 Vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19 | interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Low-dose vaccine (18-59 years) & Two dose regimen (Experimental): two doses of low-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Interventions: Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Two dose regimen
- Low-dose vaccine (18-59 years) & Three dose regimen (Experimental): three doses of low-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Interventions: Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Three dose regimen
- High-dose vaccine (18-59 years) & Two dose regimen (Experimental): two doses of high-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Interventions: Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Two dose regimen
- High-dose vaccine (18-59 years) & Three dose regimen (Experimental): three doses of high-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Interventions: Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Three dose regimen
- Low-dose vaccine (60-85 years) & Two dose regimen (Experimental): two doses of low-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Interventions: Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Two dose regimen
- Low-dose vaccine (60-85 years) & Three dose regimen (Experimental): three doses of low-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Interventions: Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Three dose regimen
- High-dose vaccine (60-85 years) & Two dose regimen (Experimental): two doses of high-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Interventions: Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Two dose regimen
- High-dose vaccine (60-85 years) & Three dose regimen (Experimental): three doses of high-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Interventions: Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Three dose regimen
- Low-dose placebo (18-59 years) & Two dose regimen (Placebo Comparator): two doses of placebo at the schedule of day 0, 21.
  Interventions: Biological: Low-dose placebo (18-59 years) & Two dose regimen
- Low-dose placebo (18-59 years) & Three dose regimen (Placebo Comparator): three doses of placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Low-dose placebo (18-59 years) & Three dose regimen
- High-dose placebo (18-59 years) & Two dose regimen (Placebo Comparator): two doses of placebo at the schedule of day 0, 21.
  Interventions: Biological: High-dose placebo (18-59 years) & Two dose regimen
- High-dose placebo (18-59 years) & Three dose regimen (Placebo Comparator): three doses of placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: High-dose placebo (18-59 years) & Three dose regimen
- Low-dose placebo (60-85 years) & Two dose regimen (Placebo Comparator): two doses of placebo at the schedule of day 0, 21.
  Interventions: Biological: Low-dose placebo (60-85 years) & Two dose regimen
- Low-dose placebo (60-85 years) & Three dose regimen (Placebo Comparator): three doses of placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Low-dose placebo (60-85 years) & Three dose regimen
- High-dose placebo (60-85 years) & Two dose regimen (Placebo Comparator): two doses of placebo at the schedule of day 0, 21.
  Interventions: Biological: High-dose placebo (60-85 years) & Two dose regimen
- High-dose placebo (60-85 years) & Three dose regimen (Placebo Comparator): three doses of placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: High-dose placebo (60-85 years) & Three dose regimen

INTERVENTIONS:
Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Two dose regimen — 18-59 years group, two doses of low-dose (20µg/0.5ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Arms: Low-dose vaccine (18-59 years) & Two dose regimen
Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Three dose regimen — 18-59 years group, three doses of low-dose (20µg/0.5ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Arms: Low-dose vaccine (18-59 years) & Three dose regimen
Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Two dose regimen — 18-59 years group, two doses of high-dose (40µg/1.0ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Arms: High-dose vaccine (18-59 years) & Two dose regimen
Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (18-59 years) & Three dose regimen — 18-59 years group, three doses of high-dose (40µg/1.0ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Arms: High-dose vaccine (18-59 years) & Three dose regimen
Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Two dose regimen — 60-85 years group, two doses of low-dose (20µg/0.5ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Arms: Low-dose vaccine (60-85 years) & Two dose regimen
Biological: Low-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Three dose regimen — 60-85 years group, three doses of low-dose (20µg/0.5ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Arms: Low-dose vaccine (60-85 years) & Three dose regimen
Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Two dose regimen — 60-85 years group, two doses of high-dose (40µg/1.0ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21.
  Arms: High-dose vaccine (60-85 years) & Two dose regimen
Biological: High-dose Recombinant COVID-19 vaccine (Sf9 cells) (60-85 years) & Three dose regimen — 60-85 years group, three doses of high-dose (40µg/1.0ml) Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 14, 28.
  Arms: High-dose vaccine (60-85 years) & Three dose regimen
Biological: Low-dose placebo (18-59 years) & Two dose regimen — 18-59 years group, two doses of placebo(0.5ml) at the schedule of day 0, 21.
  Arms: Low-dose placebo (18-59 years) & Two dose regimen
Biological: Low-dose placebo (18-59 years) & Three dose regimen — 18-59 years group, three doses of placebo(0.5ml) at the schedule of day 0, 14, 28.
  Arms: Low-dose placebo (18-59 years) & Three dose regimen
Biological: High-dose placebo (18-59 years) & Two dose regimen — 18-59 years group, two doses of placebo(1.0ml) at the schedule of day 0, 21.
  Arms: High-dose placebo (18-59 years) & Two dose regimen
Biological: High-dose placebo (18-59 years) & Three dose regimen — 18-59 years group, three doses of placebo(1.0ml) at the schedule of day 0, 14, 28.
  Arms: High-dose placebo (18-59 years) & Three dose regimen
Biological: Low-dose placebo (60-85 years) & Two dose regimen — 60-85 years group, two doses of placebo(0.5ml) at the schedule of day 0, 21.
  Arms: Low-dose placebo (60-85 years) & Two dose regimen
Biological: Low-dose placebo (60-85 years) & Three dose regimen — 60-85 years group, three doses of placebo(0.5ml) at the schedule of day 0, 14, 28.
  Arms: Low-dose placebo (60-85 years) & Three dose regimen
Biological: High-dose placebo (60-85 years) & Two dose regimen — 60-85 years group, two doses of placebo(1.0ml) at the schedule of day 0, 21.
  Arms: High-dose placebo (60-85 years) & Two dose regimen
Biological: High-dose placebo (60-85 years) & Three dose regimen — 60-85 years group, three doses of placebo(1.0ml) at the schedule of day 0, 14, 28.
  Arms: High-dose placebo (60-85 years) & Three dose regimen

SUMMARY:
This is a phase Ⅱ, single-center, randomized, double-blind, placebo-controlled study, to evaluate the immunogenicity and safety of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-60 and 60-85 years) with different immunization procedures (0, 21 days and 0, 14, 28 days) and doses (20μg/40μg).

DETAILED DESCRIPTION:
This is a phase Ⅱ, single-center, randomized, double-blind, placebo-controlled study, to evaluate the immunogenicity and safety of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-60 and 60-85 years) . The phase Ⅱ clinical trials designed 8 research group, including two immunization procedures (0, 21 days and 0, 14, 28 days), two doses (20μg/0.5ml, 40μg/1.0ml) and two ages group (adults and elder): Each group including 120 participants. Vaccination or placebo group will be randomly assigned to receive in a 5:1 ratio, 960 in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above.
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able and willing to complete all the secluded study process during the whole study follow-up period (about 7 months).
* Axillary temperature ≤37.0℃.
* General good health as established by medical history and physical examination.

Exclusion Criteria:

First dose exclusion criteria:

* Positive serum immunoglobulin M (IgM) and IgG to the SARS-CoV-2.
* A Known History of HIV infection
* Family history of seizure, epilepsy, brain or mental disease.
* Participant that has an allergic history to any ingredient of vaccines.
* Woman who is pregnant, breast-feeding or positive in pregnancy test on day of enrollment, or is planning to be pregnant during the next 6 months.
* Any acute fever disease or infections.
* Have a medical history of SARS.
* Have serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and not well-controlled.
* Major chronic illness, such as asthma, diabetes, or thyroid disease, and not well-controlled.
* Hereditary angioneurotic edema or acquired angioneurotic edema.
* Urticaria in last one year.
* Asplenia or functional asplenia.
* Platelet disorder or other bleeding disorder may cause injection contraindication.
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylactics treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months.
* Prior administration of other research medicines in last 1 month.
* Prior administration of attenuated vaccine in last 1 month.
* Prior administration of subunit vaccine or inactivated vaccine in last 14 days.
* Being treated for tuberculosis.
* Any condition that in the opinion of the investigators may interfere with the evaluation of study objectives.

Exclusion criteria for subsequent doses:

* Patients with severe allergic reactions after the previous dose of vaccination;
* Patients with serious adverse events causally related to the previous dose of vaccination.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Geometric mean (GMT) of specific antibody | 1 months after immunization in each study group
  Geometric mean (GMT) of specific antibody against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Spike protein Receptor-binding domain(S-RBD) protein (ELISA)
The incidence of adverse reaction (AR) | 0 to 7 days after vaccination in each study group
  The incidence of adverse reaction (AR)

SECONDARY OUTCOMES:
The incidence of adverse events (AE) | 0 to 28 days after vaccination in each study group
  The incidence of adverse events (AE)
The incidence of severe adverse events (SAE) | 0 to 28 days after vaccination in each study group
  The incidence of severe adverse events (SAE)
The incidence of serious adverse events | 6 months after vaccination in each study group
  The incidence of serious adverse events
Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies | 1 months after immunization in each study group
  Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies (euvirus and pseudovirus-neutralizing assays)
The positive conversion rate of S-RBD protein-specific antibody | 14 days, 30 days after immunization in each study group
  The positive conversion rate of S-RBD protein-specific antibody (ELISA) against SARS-CoV-2
Geometric mean fold increase (GMI) of S-RBD protein-specific antibody | 14 days, 30 days after immunization in each study group
  Geometric mean fold increase (GMI) of S-RBD protein-specific antibody (ELISA) against SARS-CoV-2
Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies | 14 days after immunization in each study group
  Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies (euvirus and pseudovirus-neutralizing assays)
The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody | 14 days, 30 days after immunization in each study group
  The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody (euvirus and pseudovirus neutralization test)
Geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific neutralizing antibodies | 14 days, 30 days after immunization in each study group
  Geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific neutralizing antibodies (eucivirus and pseudovirus neutralization assays)

OTHER OUTCOMES:
The consistency analysis of the specific antibody and the specific neutralizing antibody | 1 months after immunization in each study group
  The consistency analysis of the specific antibody (ELISA) and the specific neutralizing antibody (euvirus and pseudovirus neutralization assays) against SARS-CoV-2 S-RBD protein
The geometric mean titer (GMT) ratio of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody | 1 months after immunization in each study group
  The geometric mean titer (GMT) ratio of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody in each study groups
The persistence (GMT，GMI，positive conversion rate) of specific antibodies | 6 months after vaccination in each study group
  The persistence (GMT，GMI，positive conversion rate) of specific antibodies against SARS-CoV-2 S-RBD protein
Subtypes of immunoglobulin G (IgG) antibodies | 1 months after immunization in each study group
  Subtypes of IgG antibodies against the S-RBD protein of SARS-CoV-2 after immunization in each study group

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China